CLINICAL TRIAL: NCT06399952
Title: A Prospective, Longitudinal and Observational Natural History Study for Children and Adults With Baker Gordon Syndrome - Genetic Autism Alliance
Brief Title: Baker Gordon Syndrome Natural History Study
Acronym: BAGOS
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, W. David Arnold, Executive Director, UM System NextGen Precision Health Initiative Professor, Physical Medicine and Rehabilitation, University of Missouri-Columbia
Other Study IDs: 2080722; SYT1 (Registry Identifier: Synaptotagmin 1-Associated Neurodevelopmental Disorder)
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-09

CONDITIONS: Rare Diseases; Autism or Autistic Traits; Development Delay; SYT-SSX Fusion Protein Expression; Sleep Disorder; Epilepsy, Generalized; Motor Delay
Keywords: Baker Gordon Syndrome; BAGOS; Synaptotagmin 1-Associated Neurodevelopmental Disorder
MeSH Terms: conditions — Rare Diseases; Autistic Disorder; Learning Disabilities; Sleep Wake Disorders; Epilepsy, Generalized; Psychomotor Disorders | interventions — Electroencephalography; Whole Genome Sequencing; High-Throughput Nucleotide Sequencing; Inhibitory Postsynaptic Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for whole and long genome sequencing Skin fibroblasts for induced pluripotential stem cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) — Participants will undergo a 5-10 minute non-anesthesia brain MRI in order to evaluate for changes in brain structure. A 20 to 30 minutes 20 channel surface electroencephalography will be performed in the wake and sleep states.
  Other Names: Electroencephalography (EEG)
Genetic: Whole Genome Sequencing — 15 milliliters of blood will be collected at the initial visit. Blood samples will be centrifuged, and plasma stored in the University of Missouri Next Gen Precision Health building. Next generation whole genome sequencing and proteomics will be performed on plasma samples. Additional blood will be collected for the DNA biobank.
  Other Names: Next Generation Sequencing
Other: Induced Pluripotential Stem Cells — A 3 mm skin punch biopsy will be collected for developing induced pluripotential stem cells.
  Other Names: iPSP

SUMMARY:
The goal of this study is to conduct a prospective, longitudinal assessment of the natural clinical progression of children and adults with Synaptotagmin1-Associated Neurodevelopmental Disorder also known as Baker Gordon Syndrome (BAGOS). This will be performed by acquiring baseline measurements and developing effective outcome measures and diagnostic tools for the disorder, to prepare the healthcare system for future clinical trials.

DETAILED DESCRIPTION:
The current natural history study is being conducted in anticipation of future treatments for patients with confirmed BAGOS. The study is an important avenue of investigation that will increase the understanding of the disorder and lead to important diagnostic and therapeutic advances. Its purpose is to identify demographic, genetic, environmental, and treatment modalities and concomitant medications that correlate with the disease's development and outcomes. This study will use standard scales and questionnaires for the assessment of global development, language, memory, and motor function, and by collecting sleep and seizure diaries. A small blood sample will be collected for whole genome sequencing and proteomic analysis. Brain imaging (MRI) and electroencephalography (EEG) recordings will be collected to identify disease biomarkers. The investigators will also be asking participants to provide a small skin sample for the development of patient specific stem cells which will be used to further understand the impact of Synaptotagmin1 mutations on neurodevelopment and as a potential screen for future therapies.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Baker Gordon syndrome.
* 0-99 years
* Ability to send medical records and diagnostic test results.
* Ability to complete tests and questionnaires.

Exclusion Criteria:

• The presence of another condition or co-morbidity unrelated to Baker Gordon syndrome, that affects neurodevelopment.

In this study, the primary caregivers/LAR for each participant diagnosed Baker Gordon Syndrome will be also considered participants.

Caregivers/LAR will have to meet the following inclusion criteria:

* >18 years.
* Legal caregiver of the patient diagnosed with a Baker Gordon Syndrome.
* Willingness to follow study procedures, as assessed by the research team.
* Willingness to sign the consent form.
* Ability to understand all the information regarding the study, as assessed by the research team.

Caregivers/LAR Exclusion Criteria:

• Less than 18 years old.

Ages: 0 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study Population:
  * Genetically confirmed BAGOS
  * 0-99 years
  This study will comprehensively evaluate the natural clinical progression of the disease using scales and questionnaires for the assessment of motor function and global development, and by collecting sleep and seizure diaries. In addition, genetic and proteomic analysis, EEG recordings and brain MRI will be collected to identify biomarkers that will indicate disease progression or improvements following treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Collection of relevant medical data (retrospective and prospective) | 24 months
  Collection of demographic data, BAGOS-related medical history, past medical and surgical history, current medication, history of immunizations and family medical history.
Neurological Assessment Scale | 24 months
  Hammersmith Infant Neurological Examination (HINE) (0-2 years ONLY). Maximum global score of 78. Higher scores indicate a higher degree of neurological performance.
Clinical Global Impressions Scale - Practitioner | 24 months
  Scales whereby practitioner rates from 1 to 7 the overall improvement/deterioration of the participant affected by BAGOS. One is improved and 7 denotes deterioration.
Pediatric Evaluation of Disability Inventory | 24 months
  Pediatric Evaluation of Disability Inventory assesses key functional capabilities and performance in children ages 6 months to 7 years.
Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | 24 months
  The PEDI-CAT is a computer adaptive caregiver report which measures Daily Activities, Mobility, Social/Cognitive, and Responsibility. It's designed for use with children and youth with a variety of physical and/or behavioral conditions.

SECONDARY OUTCOMES:
Gross motor milestones | 24 months
  World Health Organization (WHO) Motor Milestones. Scale of 6 gross motor milestones. Lower scores denote worse motor function.
Global development assessment scale | 24 months
  Bayley Scales of Infant and Toddler Development - 4 (BSID-4) for Developmental delays. Scale is divided into five domains, which are further divided into subdomains. The first step is to calculate the starting point by beginning with the items that are age appropriate. The starting point is validated if three consecutive items are achieved. If the participant affected by Baker Gordon Syndrome does not achieve three consecutive items in a row at the age-appropriate starting point, the evaluator must go backwards to the lower age-starting point until the participant affected by Baker Gordon Syndrome achieves three items in a row. The assessment stops once five items in a row are not achieved.
Vineland Adaptive Behavior Scales Third Edition | 24 months
  Vineland Adaptive Behavior Scales Third Edition is the leading instrument for supporting the diagnosis of intellectual and developmental disabilities. Vineland-3 not only aids in diagnosis, but provides valuable information for developing educational and treatment plans
Aberrant behavior assessment (ABC) | 24 months
  Aberrant Behavior Checklist-Community (ABC-C). This scale comprises 58 items and is divided into five subdomains. The ABC-C is designed on a four-point scale with the lowest score representing less-affected patients while the highest score represents most-affected patients.
Behavior Assessment System for Children (BASC), 3rd Edition | 24 months
  Behavior Assessment System for Children (BASC), 3rd Edition. A comprehensive set of rating scales and forms, BASC-3 helps participants understand the behaviors and emotions of children and adolescents
Conners 4th Edition | 24 months
  Conners 4th Edition (Conners 4™) provides a comprehensive assessment of symptoms and impairments associated with ADHD and common co-occurring problems and disorders in children and youth aged 6 to 18 years.
Motor function assessment | 24 months
  Functional Mobility Scale (FMS). Scale which rates the walking ability in three different walking distances, and these distances will be rated on a 6-point scale. Higher scored denote less impairment.
Pediatric Sleep Questionnaire (PSQ) | 24 months
  A 22-point questionnaire that assesses the sleep patterns and potential abnormalities in children and their affected quality of life.
Test of Everyday Attention for Children 2nd Edition (TEA-Ch2) | 24 months
  Test of Everyday Attention for Children Second Edition (TEA-Ch2) uniquely measures separable aspects of attention.
NEPSY 2nd edition | 24 months
  NEPSY®-II results provide information relating to typical childhood disorders, enabling accurate diagnosis and intervention planning for success in school and at home.
The Infant/Toddler Sensory Profile | 24 months
  The Infant/Toddler Sensory Profile® was developed to evaluate sensory processing patterns in the very young. The results provide understanding of how sensory processing affects the child's daily functioning performance.
Mullen Scales of Early Learning | 24 months
  Mullen Scales of Early Learning is a developmentally integrated system that assesses language, motor, and perceptual abilities, measures cognitive ability and motor development quickly and reliability.

OTHER OUTCOMES:
Health economics | 24 months
  Interview with Caregivers
Clinical trial readiness | 24 months
  Demographic data collection
Clinical trial readiness | 24 months
  Facilities Preparation
Laboratory tests | 24 months
  Genomic and proteomic analysis of plasma samples to determine biomarkers of disease progression
Electroencephalogram activity recordings (EEG) | 24 months
  Electroencephalogram (EEG) to record brain activity of Baker Gordon Syndrome patients over a 2-hour period.
Brain magnetic resonance imaging (MRI) | 24 months
  Brain magnetic imaging (MRI) to measure the brain grey and white matter volume.

CONTACTS AND LOCATIONS:
Overall Officials: W. David Arnold, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Riggs E, Shakkour Z, Anderson CL, Carney PR. SYT1-Associated Neurodevelopmental Disorder: A Narrative Review. Children (Basel). 2022 Sep 22;9(10):1439. doi: 10.3390/children9101439. PMID 36291375
- See also: Baker Gordon Syndrome Foundation — http://www.bagosfoundation.org
- See also: University of Missouri NextGen Precision Health — https://precisionhealth.missouri.edu
- See also: Thompson Center for Autism and Neurodevelopment — https://precisionhealth.missouri.edu